CLINICAL TRIAL: NCT06542757
Title: Evaluation of Tumor Control Based on Serial Multiparametric MRI and Post-Treatment Biopsies For Patients Treated With Dose Intensification to the Dominant Intra-Prostatic Lesion (DIL) Using Ultra-Hypofractionated, MR-Guided Radiotherapy (TUMORNATOR I)
Brief Title: Evaluation of Tumor Control Based on Serial Multiparametric MRI and Post-Treatment Biopsies For Patients Treated With Dose Intensification to the Dominant Intra-Prostatic Lesion (DIL) Using Ultra-Hypofractionated, MR-Guided Radiotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-01590
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer
Keywords: intensity-modulated radiotherapy; MR-guided
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- MRI-guided Intensity Modulated Radiotherapy (Experimental): All patients will undergo the injection of a hydrogel rectal spacer (SpaceOAR) 1 week before simulation. Patients will undergo ultra-hypofractionated radiation utilizing MR-guided, daily online adaptive planning. Patients will receive 9 Gy/fraction for five fractions for a total dose of 45 Gy to the prostate DIL while the rest of the prostate will be treated to a minimum dose to the rest of the prostate of 30 Gy in five fractions. Radiation will be given every other day, Monday through Friday, until 5 treatments have been completed. Patients will be followed at three and six months after treatment, and every six months thereafter through month 24 (+/- 4 weeks).
  Interventions: Radiation: 1.5 T Elekta Unity MR-Linac system; Device: Hydrogel rectal spacer (SpaceOAR)

INTERVENTIONS:
Radiation: 1.5 T Elekta Unity MR-Linac system — Patients will receive 9 Gy/fraction (45 Gy total) for five fractions to the DIL, while the remainder of the prostate will be treated to 30 Gy in 5 fractions.
Device: Hydrogel rectal spacer (SpaceOAR) — A rectal spacer will be placed one week prior to simulation to achieve a separation of approximately 1 cm between the prostate and anterior rectal wall to further minimize rectal toxicity in these patients. The hydrogel will remain in the body for about 12 weeks.

SUMMARY:
The purpose of this study is to assess the impact of this MR-guided radiotherapy on tumor control of the dominant intraprostatic lesion among patients with intermediate risk prostate cancer. This study of Radiotherapy to the Prostate and Dominant Lesion Using Ultra-Hypofractionated, MR-adaptive Radiation Therapy aims to evaluate tumor control after definitive ultra-hypofractionated external beam radiation therapy (including a simultaneously delivered high-dose boost to a dominant lesion as detected on prostate magnetic resonance imaging (MRI)) in patients with intermediate-risk prostate cancer. This will incorporate the use of multiparametric MRI for target segmentation and the use of the MR-linac with adaptive radiation planning to treat the prostate gland, incorporating a dose boost to the dominant intraprostatic lesion (DIL) that is visible on T2-weighted and diffusion-weighted imaging and de-escalation of dose to the remainder of the prostate.

ELIGIBILITY:
Inclusion Criteria:

1. Intermediate-risk prostate cancer patients will be eligible for this study. Risk groups will be assigned as per National Comprehensive Cancer Network (NCCN) guidelines. Intermediate-risk patients will be defined as:

   * PSA 10-20 ng/ml or
   * Gleason score = 7 or
   * Clinical stage T2b/T2c (T2b: the tumor has spread to more than one-half of one side of the prostate, but not to both sides. T2c: the cancer has invaded both sides of the prostate)
2. Age > 18
3. Karnofsky Performance Status (KPS) > 80
4. Prostate size < 90 cc
5. Presence of a T2-visible prostatic lesion with maximum dimension of ≥ 0.5 cm and no more than two additional disease foci with a documented Prostate Imaging Reporting and Data System (PIRADS) 4-5 lesion
6. MRI findings: Lesion may contact the capsular edge, possible extracapsular extension (ECE) permitted
7. International Prostate Symptom Score < 18
8. Satisfy all MRI screening criteria and be willing to fill out the standard MRI screening form

Exclusion Criteria:

1. Gleason score >7
2. PSA >20 ng/mL
3. Prior or concurrent androgen deprivation therapy for prostate cancer
4. MRI findings: suspicious for/probable ECE
5. MRI findings: >2 disease foci identifiable
6. Evidence of metastatic disease on bone scan or MRI/CT
7. MRI ineligibility due to: the presence of a cardiac pacemaker, defibrillator, or other implanted metallic or electronic device which is considered MR unsafe; severe claustrophobia; inability to lie flat for the duration of the study; etc.
8. Metallic implant or device in the pelvis that might distort the local magnetic field and compromise quality of mp-MRI
9. Lateral pelvic separation greater than 50 cm and/or anterior-posterior separation greater than 35 cm which are incompatible with MR for Calculating ATtenuation (MRCAT) reconstruction
10. Contra-indications to receiving gadolinium contrast
11. KPS < 80
12. Pelvic or Prostate MRI or CT (MRI preferred) evidence of radiographic T3, T4, or N1 disease
13. Prior history of transurethral resection of the prostate
14. Prior history of urethral stricture
15. Prior history of pelvic irradiation
16. History of inflammatory bowel disease
17. Unable to give informed consent
18. Unable to complete quality of life questionnaires
19. Abnormal complete blood count, including any of the following:

    * Platelet count less than 75,000/ml
    * Hb level less than 10 gm/dl
    * White blood cell (WBC) less than 3.5/ml
    * Abnormal renal function tests (creatinine > 1.5)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Negative biopsy rate 24 months post-treatment | 24 months post-treatment
  Outcome measure will be assessed via repeat biopsy of the dominant lesion as seen on mp-MRI
Serious toxicity rate 24 months post-treatment | 24 months post-treatment
  Outcome measure will be assessed using NCI CTCAE v5.0 for gastrointestinal and genitourinary toxicity.

SECONDARY OUTCOMES:
Prostate Specific Antigen (PSA) relapse rate at 24 months post-treatment | 24 months post-treatment
Proportion of patients with radiation-induced response in the dominant prostatic lesion 6 months post treatment | 6 months post-treatment
  Outcome measure will be assessed using multi-parametric MR imaging.
Proportion of patients with radiation-induced response in the dominant prostatic lesion 24 months post treatment | 24 months post-treatment
  Outcome measure will be assessed using multi-parametric MR imaging.
Change in International Prostate Symptom Score (I-PSS) | Baseline, Month 3
  The I-PSS is based on the answers to seven questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic). Score are classified as follows: 0 - 7 = mildly symptomatic; 8 - 19 = moderately symptomatic; 20 - 35 = severely symptomatic.
Change in International Prostate Symptom Score (I-PSS) | Baseline, Month 6
  The I-PSS is based on the answers to seven questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic). Score are classified as follows: 0 - 7 = mildly symptomatic; 8 - 19 = moderately symptomatic; 20 - 35 = severely symptomatic.
Change in International Prostate Symptom Score (I-PSS) | Baseline, Month 12-18
  The I-PSS is based on the answers to seven questions concerning urinary symptoms. Each question is assigned points from 0 to 5 indicating increasing severity of the particular symptom. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic). Score are classified as follows: 0 - 7 = mildly symptomatic; 8 - 19 = moderately symptomatic; 20 - 35 = severely symptomatic.
Change in International Index of Erectile Function (IIEF) score | Baseline, Month 3
  The IIEF consists of 11 items, grouped into five factors: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. Items are scored in a 1-5 Likert-type scale, with higher scores indicating better erectile function. Erectile dysfunction (ED) severity is classified into five categories: no ED (score 22-25), mild (17-21), mild to moderate (12-16), moderate (8-11), and severe (5-7).
Change in International Index of Erectile Function (IIEF) score | Baseline, Month 6
  The IIEF consists of 11 items, grouped into five factors: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. Items are scored in a 1-5 Likert-type scale, with higher scores indicating better erectile function. ED severity is classified into five categories: no ED (score 22-25), mild (17-21), mild to moderate (12-16), moderate (8-11), and severe (5-7).
Change in International Index of Erectile Function (IIEF) score | Baseline, Month 12-18
  The IIEF consists of 11 items, grouped into five factors: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. Items are scored in a 1-5 Likert-type scale, with higher scores indicating better erectile function. ED severity is classified into five categories: no ED (score 22-25), mild (17-21), mild to moderate (12-16), moderate (8-11), and severe (5-7).
Change in genomic classifier (GC) Decipher score | Baseline, 6 months post-treatment
  Scores are derived from the expression of 22 genes. Decipher scores are a continuous variable reported on a scale of 0 to 1. These scores are then stratified to three risk-categories: low (<0.45), intermediate (≥ 0.45 - < 0.6) and high (≥ 0.6)
Change in GC Decipher score | Baseline, 24 months post-treatment
  Scores are derived from the expression of 22 genes. Decipher scores are a continuous variable reported on a scale of 0 to 1. These scores are then stratified to three risk-categories: low (<0.45), intermediate (≥ 0.45 - < 0.6) and high (≥ 0.6)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zelefsky, M.D, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared to achieve aims in the approved proposal beginning 3 months and ending 5 years following article publication provided the researchers who provide a methodologically sound proposal executes a data use agreement with NYU Langone Health. Requests may be directed to: Michael.Zelefsky@nyulangone.org. The protocol, statistical analysis plan, informed consent form, and clinical study report will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal will be provided access to achieve aims in the approved proposal. Requests should be directed to Michael.Zelefsky@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.